CLINICAL TRIAL: NCT07054268
Title: Nurse-Led Implementation of the ABCDEF Bundle: Evidence-Based Strategies for ICU Delirium Management
Brief Title: Nurse-Led Implementation of the ABCDEF Bundle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Alaa Eldin Moustafa Hamed, Lecturer of Psychiatric and mental health Nursing, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NURSERC2023/12/10
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-03

CONDITIONS: Delirium in the Intensive Care Unit
Keywords: ICU delirium; evidence-based nursing; nursing interventions; critical care; patient outcomes.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The study group received a nurse-led implementation of the ABCDEF bundle, which included structured interventions to assess and manage pain, conduct spontaneous awakening and breathing trials, optimize sedation choices, screen for and manage delirium, promote early mobility, and engage family members. ICU nurses delivered the intervention following standardized protocols to ensure consistency and adherence to the bundle components.
  Interventions: Other: Nurse-Led ABCDEF Bundle Implementation
- control group (No Intervention): The control group received standard ICU care as per the hospital's existing protocols. No structured implementation of the ABCDEF bundle was applied, and nursing care followed routine clinical practices without specific emphasis on coordinated bundle elements.

INTERVENTIONS:
Other: Nurse-Led ABCDEF Bundle Implementation — This intervention is distinguished by its structured, nurse-led delivery of all six components of the ABCDEF bundle, with nurses serving as primary implementers rather than multidisciplinary teams. Unlike other studies that may focus on select elements of the bundle or physician-led application, this study emphasizes standardized nursing protocols and daily documentation to ensure consistent implementation and evaluation across all components specifically targeting delirium prevention and management in ICU patients.
  Arms: Study Group

SUMMARY:
This study evaluated the effectiveness of a nurse-led implementation of the ABCDEF bundle, an evidence-based, interprofessional care framework, in the prevention and management of delirium among Intensive Care Unit (ICU) patients. The intervention aimed to reduce the incidence and severity of ICU delirium, decrease agitation, and improve patient outcomes through structured nursing interventions guided by the ABCDEF approach.

DETAILED DESCRIPTION:
The study employed a single-center, quasi-experimental clinical design with two parallel groups: an intervention group that received the nurse-led ABCDEF bundle and a control group that received standard ICU care. No randomization was applied, but baseline characteristics were matched where possible to control for confounding variables.

The study was conducted in the adult ICU of a tertiary care hospital. Eligible participants included adult patients (≥18 years) who were admitted to the ICU with an expected stay of at least 48 hours. Patients with pre-existing cognitive impairment, severe neurological damage, or those in a persistent vegetative state were excluded.

The intervention group received structured nursing care guided by the ABCDEF bundle, delivered by trained ICU nurses. The protocol included routine pain assessments and management strategies; daily spontaneous awakening and breathing trials; evidence-based sedation choices minimizing benzodiazepine use; systematic delirium screening using a validated tool (e.g., ICDSC); early mobilization practices appropriate to the patient's clinical status; and inclusion of family members in care planning and education.

The control group received usual ICU care without the formal implementation of the ABCDEF bundle.

The primary outcome was the incidence of delirium during the ICU stay, measured using a validated tool (e.g., ICDSC or CAM-ICU). Secondary outcomes included agitation levels, duration of delirium episodes, ICU length of stay, adherence to individual ABCDEF components, use of physical restraints, and sedative/analgesic dosages.

Data were collected prospectively from patient medical records, bedside observations, and standardized assessment tools. Daily monitoring was conducted to ensure fidelity to the intervention and accurate documentation of outcomes.

Ethical approval was obtained from the institutional review board. Written informed consent was obtained from patients or their legal representatives where applicable.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill adult patients aged 18 years or older
* Admitted to the ICU at Ain Shams University Hospitals within 48 hours of enrollment
* Clinically stable to undergo assessment and nursing intervention
* Able to provide informed consent personally or via a legally authorized representative
* Both male and female patients included

Exclusion Criteria:

* Documented cognitive impairment or pre-existing psychiatric illness
* Severe neurological conditions (e.g., advanced stroke, traumatic brain injury)
* Deep sedation level (Richmond Agitation-Sedation Scale [RASS] score < -4)
* Terminal illness requiring palliative or end-of-life care
* Patients who declined participation or did not meet eligibility screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of ICU Delirium | From ICU admission to ICU discharge or up to 7 days, whichever occurs first
  The presence or absence of delirium will be assessed daily using the Intensive Care Delirium Screening Checklist (ICDSC), a validated tool. Delirium is defined as an ICDSC score ≥4. The outcome will measure the proportion of patients who develop delirium during their ICU stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided